CLINICAL TRIAL: NCT06314373
Title: A Phase I/II Study to Assess the Safety, Tolerability, PK/PD, and Preliminary Efficacy of HSK39775 Tablet Monotherapy in Participants With Advanced Solid Malignancies
Brief Title: A Study for HSK39775 in Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xizang Haisco Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK39775-101/201
Record Dates: First submitted 2024-02-29; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose Escalation:Participants will receive escalating doses of HSK39775
  Interventions: Drug: HSK39775 Monotherapy
- Cohort Expansion (Experimental): Cohort Expansion:Participants will receive HSK39775 at the identified RP2D
  Interventions: Drug: HSK39775 Monotherapy

INTERVENTIONS:
Drug: HSK39775 Monotherapy — HSK39775 will be administered orally once daily

SUMMARY:
This research is designed to determine if HSK39775 is safe, tolerable, and has anti-cancer activity in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at screening
2. Histological or cytological confirmation of advanced malignancy, have failed or intolerant to the standard-of-care treatment or no standard therapy is recognized or standard therapy is unavailable
3. Eastern Cooperative Oncology Group performance status 0 or 1
4. Patients must have evaluable disease as defined
5. Life expectancy of ≥ 12 weeks
6. Adequate organ and bone marrow function per protocol
7. Female patients who are women of childbearing potential with confirmed of a negative pregnancy test within 7 days prior to the first dose and agreement to the use of effective contraceptive method at the same time during study treatment period and for up to 6 months after the last dose of study treatment. Male patients must be willing to use effective contraception during the study treatment period and for up to 6 months after the last dose of study treatment
8. Written informed consent must be obtained

Exclusion Criteria:

1. Known allergies to HSK39775 or its excipients
2. Prior anticancer treatment is ineligible per protocol
3. Subjects who have had continuous corticosteroids at a dose of >10 mg prednisone/day or equivalent within 4 weeks prior to the first dose of study treatment
4. Subjects who have had live vaccine within 4 weeks prior the first dose of study treatment
5. Currently participating in a study of another investigational agent or device
6. Subjects who have had received another agent with same target
7. Subjects who have not recovered (to grade ≤1 or baseline) from toxicities related to prior therapies
8. Subjects who have had received drugs that may have drug-drug interaction potential within 4 weeks or 5 half-lives prior to the first dose of study treatment
9. Subjects who have had received major surgery within 4 weeks prior the first dose of study treatment
10. Central nervous system metastases associated with neurological symptoms
11. Active hepatitis B or hepatitis C infection
12. A history of immunodeficiency
13. Clinically relevant cardiovascular disease as delined by protocol
14. Inability to swallow the formulated product or impairment of GI function or disease that may significantly alter the absorption of study drug
15. A female patient who is pregnant or lactating
16. Other conditions, in investigator's opinion, not suitable to participate in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
AE/SAE | From time of informed consent to 28 days post last dose or start of other anti-cancer therapies
  Safety data
DLT | From the start of first dose to the end of Cycle1(each cycle is 28 days)
  Safety data
MTD/MAD | From the start of first dose to the end of Cycle1(each cycle is 28 days)
  Safety data

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | At predefined intervals throughout the treatment period(approximately 12 weeks)
Area Under Curve[AUC] | At predefined intervals throughout the treatment period(approximately 12 weeks)
Time to maximum observed concentration [Tmax] | At predefined intervals throughout the treatment period(approximately 12 weeks)
Elimination half-life [t1/2] | At predefined intervals throughout the treatment period(approximately 12 weeks)
Overall Response Rate (ORR) per RECIST V1.1 | From Screening to confirmed progressive disease or date of death from any cause, whichever came first[approximately 1 year]
Progression Free Survival | From Screening to confirmed progressive disease or date of death from any cause, whichever came first[approximately 1 year]
Time To Response | From Screening to confirmed progressive disease or date of death from any cause, whichever came first[approximately 1 year]
Disease Control Rate | From Screening to confirmed progressive disease or date of death from any cause, whichever came first[approximately 1 year]
Best percentage change in target lesion | From Screening to confirmed progressive disease or date of death from any cause, whichever came first[approximately 1 year]

CONTACTS AND LOCATIONS:
Locations (1):
- Fundan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No